CLINICAL TRIAL: NCT02129270
Title: Phase 4 Study of Hematoma Block for Reduction of Distal Radius Fractures
Brief Title: Hematoma Block for Reduction of Distal Radius Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 158-13-EMC
Record Dates: First submitted 2014-04-07; First posted 2014-05-02 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Fractures of the Distal Radius
Keywords: Fractures of the distal radius; Hematoma block; Lidocaine

ARMS (2):
- Lidocaine HCl 2% (Active Comparator): Lidocaine HCl 2% (200mg/10ml) 10 ml.
  Interventions: Drug: Lidocaine HCl 2% .
- Lidocaine HCl 1% (Experimental): Lidocaine HCl 1% (100mg/10ml) 15-20 ml.
  Interventions: Drug: Lidocaine HCl 1%

INTERVENTIONS:
Drug: Lidocaine HCl 2% . — comparison of different dosages of drug
  Other Names: ESRACAIN
  Arms: Lidocaine HCl 2%
Drug: Lidocaine HCl 1% — comparison of different dosages of drug
  Other Names: ESRACAIN
  Arms: Lidocaine HCl 1%

SUMMARY:
The purpose of this study is to Prove that injection of 15 to 20 mL of lidocaine 1% into the fracture site (Hematoma block) is more effective in terms of pain relieving then injection of 10 mL of lidocaine 2%, and equally safe in terms of complications, for closed reduction of distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Fractures of the distal radius, with or without ulna fracture

Exclusion Criteria:

* Children,
* pregnant women,
* patients with infection or suspected infection on the site for injection.
* Patients whose condition requires general anesthesia (patients with more fractures other than the distal radius and ulna, patients with many damage...)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
This study will be measured effective in terms of pain relieving with Visual Analog Scale. | 1 year

SECONDARY OUTCOMES:
This study will be measured safe in terms of complications to injection. | 1 year
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Nimrod Rozen, Prof., Principal Investigator — HaEemek Medical Center
Locations (1):
- HaEmek medical center, Afula, Israel